CLINICAL TRIAL: NCT06485921
Title: Comparison of the Effectiveness of Ischemic Compression and Instrument Assisted Soft Tissue Mobilization on Pain and Function in Patients With Nonspecific Neck Pain
Brief Title: Comparison of Two Treatments on Nonspecific Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mouna Khosravi, Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUC-FTR-MK-01
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain
Keywords: Neck pain; Trigger point; Exercise; Physical therapy; Manual therapy
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Acupressure; Exercise

STUDY DESIGN:
Intervention Model Description: Three groups with conventional therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ischemic compression GROUP (Active Comparator): This group will receive 90 seconds of ischemic compression on myofascial trigger points in the trapezius, levator scapulae, supraspinatus, infraspinatus, and splenius cervicis, along with exercises and suggestions for workplace modifications.
  Interventions: Other: Ischemic compression; Other: Exercise and workplace modifications
- Instrument assisted soft tissue mobilization Group (Active Comparator): This group will receive 40 seconds of sweeping and 60 seconds of swiveling by instrument-assisted soft tissue mobilization on myofascial trigger points in the trapezius, levator scapulae, supraspinatus, infraspinatus, and splenius cervicis muscles, along with exercises and suggestions for workplace modifications.
  Interventions: Other: Instrument assisted soft tissue mobilization Group; Other: Exercise and workplace modifications
- Control Group (Experimental): This group will only receive exercises and suggestions for workplace modifications.
  Interventions: Other: Exercise and workplace modifications

INTERVENTIONS:
Other: Ischemic compression — Participants will received a total of 12 treatment sessions over 6 weeks, with 2 sessions per week.
  Arms: Ischemic compression GROUP
Other: Instrument assisted soft tissue mobilization Group — Participants will received a total of 12 treatment sessions over 6 weeks, with 2 sessions per week.
  Arms: Instrument assisted soft tissue mobilization Group
Other: Exercise and workplace modifications — Participants will receive stretching and strengthening exercises for neck and scapular stabilizer muscles as a 6-week home program.

SUMMARY:
The purpose of this study was to evaluate the impact of Ischemic Compression (IC) and Instrument Assisted Soft Tissue Mobilization (IASTM) on pain, functionality, cervical range of motion, pressure pain threshold, and quality of life in patients suffering from nonspecific neck pain.

DETAILED DESCRIPTION:
Chronic nonspecific neck pain affects approximately 67% of the global population at least once in their lifetime. This type of neck pain, which is not linked to any specific cause or disease but often associated with the musculoskeletal system, can result from muscle strain or spasms in the neck. It causes functional limitations and decreases quality of life for those affected. Individuals frequently turn to healthcare services and pain-relieving medications in their efforts to manage this discomfort. Chronic nonspecific neck pain is recognized as a significant public health challenge due to its considerable socioeconomic impact. Several studies have indicated that myofascial trigger points in the neck region are associated with nonspecific neck pain and that myofascial trigger point therapy can reduce pain. Therefore, the role of myofascial trigger point therapy in the treatment of nonspecific neck pain has been emphasized in studies.

ELIGIBILITY:
Inclusion Criteria:

1. Having nonspecific neck pain and at least 3 myofascial trigger points in the back and neck muscles,
2. Pain duration exceeding 3 months,
3. Working with a computer for at least 20 hours per week for at least 1 year,
4. Pain intensity rated as at least 3 on the Visual Analog Scale (VAS),
5. Age between 18 and 50 years

Exclusion Criteria:

1. Use of anti-inflammatory, analgesic, anticoagulant, muscle relaxant, or antidepressant medications at the start of the study or within 1 week prior to the study,
2. History of cervical spine surgery or trauma,
3. Neck pain, including inflammatory rheumatic diseases,
4. Malignancy or structural deformity,
5. Coagulation disorders,
6. Presence of cervical radiculopathy or myelopathy,
7. Individuals who have undergone any physical therapy and rehabilitation interventions to the neck and back regions in the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | Six weeks
  VAS is a measurement tool commonly used to assess the intensity of pain or other symptoms. It consists of a horizontal line labeled with descriptive anchors at each end (e.g., 'no pain' to 'worst pain imaginable'). Patients mark on the line to indicate their subjective perception of symptom severity, with the distance from the starting point to the mark providing a quantitative measure. As the value on the scale increases, the perceived pain or symptom intensity also increases
Neck Disability Index (NDI) | Six weeks
  NDI is a measurement tool used to assess functional limitations in the neck region. It is commonly employed in individuals experiencing neck pain to evaluate the extent of restrictions in daily activities. NDI allows patients to subjectively assess how much their neck pain affects their daily lives. The score on the scale indicates the degree of functional impairment experienced by the patient and is used to evaluate treatment outcomes. When the score decreases, it indicates a reduction in limitations.

SECONDARY OUTCOMES:
The Work Role Functioning Questionnaire (WRFQ) | Six weeks
  WRFQ evaluates functionality and work capacity by assessing individuals' roles and functions in the workplace. It covers aspects such as work performance, job retention, and job-related functionality. The questionnaire identifies both constraints and strengths in the workplace, offering insights into employees' perceptions of their job performance and role. It is widely used to assess return to work readiness and overall work ability, with higher scores indicating improved work performance.
Cervical range of motion | Six weeks
  Individuals' active cervical range of motion includes flexion, extension, right-left lateral flexion, and rotation will measured with a universal goniometer.
Pain pressure threshold | Six weeks
  The pressure algometer (model: JTECH USA Commander) will be applied perpendicularly to the trigger point. Participants will be instructed to report the onset of discomfort. Compression will be halted upon their report, and the measurement displayed on the algometer screen will be documented. Three readings will be taken with a 30-second interval between each trial, and the average value will be recorded for analysis.
SF- 12 quality of life | Six weeks
  SF-12 Quality of Life (SF-12 QoL) is a standardized survey tool used to measure health-related quality of life in individuals. It consists of 12 questions that assess physical and mental health, daily functioning, emotional well-being, and overall perception of health status. The survey provides scores for physical and mental health components, reflecting the individual's perceived quality of life across these domains. SF-12 QoL is widely used in research and clinical settings to evaluate health outcomes, monitor changes in health status over time, and assess the impact of interventions on quality of life.
Global Rating of Change (GROC) | Six weeks
  The satisfaction levels of the participants will be evaluated using the 5-point GROC scale at the end of 6 weeks. The scale ranges from -2 to +2, where -2 indicates "I am much worse," -1 indicates "I am worse," 0 indicates "I am the same," +1 indicates "I am better," and +2 indicates "I am much better."

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Khosravi, MSc, Principal Investigator — aculty of Health Sciences, Istanbul University-Cerrahpasa, Büyükçekmece/Istanbul, Turkey
Locations (1):
- Faculty of Health Sciences, Istanbul University-Cerrahpasa, Istanbul, Büyükçekmece, Turkey (Türkiye)